CLINICAL TRIAL: NCT00868218
Title: Preparing for an Influenza Pandemic: A Phase I Study of a Parenterally Administered H5N1 Influenza Vaccine in Healthy Adults
Brief Title: Study of a Parenterally Administered H5N1 Influenza Vaccine in Healthy Adults
Acronym: PANFLUVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rebecca Cox (Other)
Collaborators: Haukeland University Hospital (Other); European Commission (Other)
Responsible Party: Sponsor-Investigator, Rebecca Cox, Professor, University of Bergen
Organization: University of Bergen (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: PANFLUVAC-2008, Version 2; EU PANFLUVAC 44115
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Influenza; Healthy
Keywords: Influenza A; pandemic; vaccine; immunogenicity; Virus; H5N1
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 30µg HA vaccine Intramuscularly administered
  Interventions: Biological: Influenza vaccine
- 2 (Active Comparator): 1.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
  Interventions: Biological: Influenza vaccine
- 3 (Active Comparator): 7.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
  Interventions: Biological: Influenza vaccine
- 4 (Active Comparator): 30µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Influenza virus strain:
  avian influenza Influenza A/Vietnam/1194/2004 NIBRG-14

SUMMARY:
The safety and tolerability of the pandemic A/H5N1 virosomal vaccine formulated with or without the 3rd generation ISCOM™ adjuvant for parenteral administration will be investigated locally and systemically and by using haematological, biochemical and immunological screening tests. The immunogenicity of the H5N1 vaccine will be assessed through the induction of local and systemic antibody and cellular immune responses. In a pandemic situation, an important aspect is the rapidity of the immune response to the H5N1 vaccine so the detailed kinetics of the immune response will be investigated. The capacity of the vaccine to elicit long lasting immunity and cross reactive immunity to H5 viruses will also be evaluated. Furthermore, the quality of the immune response induced by the vaccine will be studied. The vaccine will be administered as twice the normal human dose (30μg HA) with and without adjuvant, and in a dose sparing manor of half (7.5μg HA) and one tenth (1.5μg HA) of the normal human dose with adjuvant. Sixty subjects will receive two doses of virosomal H5N1 influenza vaccine (separated by 21 ± 4 days) by intramuscular injection into the deltoid muscle. Escalating doses will be separated by a period of one week. Four groups each containing 15 subjects will receive two doses of the pandemic virosomal A/H5N1 influenza vaccine containing:

Group 1 30µg HA IM, Group 2 1.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ IM, Group 3 7.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ IM, Group 4 30µg HA adjuvanted with 50µg 3rd generation ISCOM™ IM.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (as concluded from the medical history, physical examination, and clinical judgment) aged 19 to 50 years old
* Females using a reliable method of contraception (from 4 weeks prior to the first vaccination until 4 weeks after the second vaccination) and a negative urine pregnancy test will be required before administration of each dose of vaccine
* Signed informed consent
* Subjects able to understand and comply with the study protocol and complete the Adverse Event Form
* Subjects able to attend the scheduled visits
* Subjects with normal pre-screening values. If a subjects prescreening samples lie outside the reference values he/she will only be included in the study based upon the medical evaluation of the clinical investigator

Exclusion Criteria:

* Persons with a history of anaphylaxis or serious reactions to any vaccine
* Persons with known hypersensitivity to any of the vaccine components
* Persons who have had a temperature >38oC during the previous 72 hours
* Persons who have had an acute respiratory infection during the last 7 days
* Women who are pregnant or breast-feeding
* Persons with chronic illness at any stage that could interfere with trial conduct or compliance
* Persons who have received blood products or immunoglobulins parenterally during the previous 3 months
* Persons who have been vaccinated with any vaccine during the 4 weeks preceding the first trial vaccination
* Persons with known or suspected immunosuppressive disease or who use systemic immunosuppressive drugs
* Persons taking immunostimulant therapy
* Persons involved in another clinical trial during the last month.
* Suspected non-compliance

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haakon Sjursen, MD, Study Director — Haukeland Univeristy Hospital
Locations (1):
- Haukeland Univeristy Hospital, Bergen, Norway

REFERENCES:
- [Result] Pedersen GK, Madhun AS, Breakwell L, Hoschler K, Sjursen H, Pathirana RD, Goudsmit J, Cox RJ. T-helper 1 cells elicited by H5N1 vaccination predict seroprotection. J Infect Dis. 2012 Jul 15;206(2):158-66. doi: 10.1093/infdis/jis330. Epub 2012 May 2. PMID 22551811
- [Result] Cox RJ, Pedersen G, Madhun AS, Svindland S, Saevik M, Breakwell L, Hoschler K, Willemsen M, Campitelli L, Nostbakken JK, Weverling GJ, Klap J, McCullough KC, Zambon M, Kompier R, Sjursen H. Evaluation of a virosomal H5N1 vaccine formulated with Matrix M adjuvant in a phase I clinical trial. Vaccine. 2011 Oct 19;29(45):8049-59. doi: 10.1016/j.vaccine.2011.08.042. Epub 2011 Aug 22. PMID 21864624
- [Result] Pedersen GK, Sjursen H, Nostbakken JK, Jul-Larsen A, Hoschler K, Cox RJ. Matrix M(TM) adjuvanted virosomal H5N1 vaccine induces balanced Th1/Th2 CD4(+) T cell responses in man. Hum Vaccin Immunother. 2014;10(8):2408-16. doi: 10.4161/hv.29583. PMID 25424948
- [Result] Pedersen GK, Hoschler K, Oie Solbak SM, Bredholt G, Pathirana RD, Afsar A, Breakwell L, Nostbakken JK, Raae AJ, Brokstad KA, Sjursen H, Zambon M, Cox RJ. Serum IgG titres, but not avidity, correlates with neutralizing antibody response after H5N1 vaccination. Vaccine. 2014 Jul 31;32(35):4550-4557. doi: 10.1016/j.vaccine.2014.06.009. Epub 2014 Jun 18. PMID 24950357
- [Result] Cox RJ, Major D, Pedersen G, Pathirana RD, Hoschler K, Guilfoyle K, Roseby S, Bredholt G, Assmus J, Breakwell L, Campitelli L, Sjursen H. Matrix M H5N1 Vaccine Induces Cross-H5 Clade Humoral Immune Responses in a Randomized Clinical Trial and Provides Protection from Highly Pathogenic Influenza Challenge in Ferrets. PLoS One. 2015 Jul 6;10(7):e0131652. doi: 10.1371/journal.pone.0131652. eCollection 2015. PMID 26147369
- [Result] Nachbagauer R, Wohlbold TJ, Hirsh A, Hai R, Sjursen H, Palese P, Cox RJ, Krammer F. Induction of broadly reactive anti-hemagglutinin stalk antibodies by an H5N1 vaccine in humans. J Virol. 2014 Nov;88(22):13260-8. doi: 10.1128/JVI.02133-14. Epub 2014 Sep 10. PMID 25210189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Haukeland University hospital recrutiment in 2009
Pre-assignment Details: Haelthy person were randomly assigned to one of 4 vaccine groups
Groups:
- 30µg HA Vaccine: 30µg HA vaccine Intramuscularly administered Influenza vaccine: Influenza virus strain: avian influenza Influenza A/Vietnam/1194/2004 NIBRG-14
- 1.5µg HA Adjuvanted: 1.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
  Influenza vaccine: Influenza virus strain:
  avian influenza Influenza A/Vietnam/1194/2004 NIBRG-14
- 7.5µg HA Adjuvanted: 7.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
  Influenza vaccine: Influenza virus strain:
  avian influenza Influenza A/Vietnam/1194/2004 NIBRG-14
- 30µg HA Adjuvanted: 30µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
  Influenza vaccine: Influenza virus strain:
  avian influenza Influenza A/Vietnam/1194/2004 NIBRG-14
Period: Overall Study
Arm/Group | 30µg HA Vaccine | 1.5µg HA Adjuvanted | 7.5µg HA Adjuvanted | 30µg HA Adjuvanted
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy adults willing to join phase I trial
Groups:
- Total: Total of all reporting groups
Arm/Group | 30µg HA Vaccine | 1.5µg HA Adjuvanted | 7.5µg HA Adjuvanted | 30µg HA Adjuvanted | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [21 to 41] | 29 [21 to 44] | 31 [22 to 42] | 31 [21 to 49] | 31 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 8 | 11 | 38
  Male | 6 | 5 | 7 | 4 | 22
Region of Enrollment [Number; unit: participants]
  Norway | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Solicted Adverse Events
Description: The primary endpoints of the trial are the local and systemic adverse events and tolerability of parenterally administered virosomal H5N1 influenza vaccine with or without 3rd generation ISCOM™ adjuvant.
Time Frame: three months
Measure: Number; unit: participants
Arm/Group | 30µg HA Vaccine | 1.5µg HA Adjuvanted | 7.5µg HA Adjuvanted | 30µg HA Adjuvanted
Number analyzed (Participants) | 15 | 15 | 15 | 15
participants | 8 | 12 | 13 | 14

2. Primary Outcome: Adverse Events
Time Frame: 42 days
Measure: Number; unit: participants
Groups:
- 1.5µg HA Adjuvanted: 1.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
- 30µg HA Vaccine: 30µg HA vaccine Intramuscularly administered
- 7.5µg HA Adjuvanted: 7.5µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
- 30µg HA Adjuvanted: 30µg HA adjuvanted with 50µg 3rd generation ISCOM™ Intramuscularly administered
Arm/Group | 1.5µg HA Adjuvanted | 30µg HA Vaccine | 7.5µg HA Adjuvanted | 30µg HA Adjuvanted
Number analyzed (Participants) | 15 | 15 | 15 | 15
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Immunogenicity of a Non-adjuvanted and 3rd Generation ISCOM™ Adjuvanted Virosomal H5N1 Influenza Vaccine
Description: Number of participants with haemagglutination inhibition tigers >= 32 at the long term time point (1 year post vaccination).
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | 1.5µg HA Adjuvanted | 30µg HA Vaccine | 7.5µg HA Adjuvanted | 30µg HA Adjuvanted
Number analyzed (Participants) | 15 | 15 | 15 | 15
participants | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: AE were solicited for 42 days after vaccination
Description: Each participant received an AE form which was returned to the clinic 21 days after each vaccination.
Arm/Group | 30µg HA Vaccine | 1.5µg HA Adjuvanted | 7.5µg HA Adjuvanted | 30µg HA Adjuvanted
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 8/15 | 13/15 | 12/15 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30µg HA Vaccine (N=15) | 1.5µg HA Adjuvanted (N=15) | 7.5µg HA Adjuvanted (N=15) | 30µg HA Adjuvanted (N=15)
local or systemic reactions (Infections and infestations) | 8 (8) | 13 (13) | 12 (12) | 13 (13) — Local: redness, local itching, oedema/local swelling, pain at the injection site, ecchymosis, hardness/induration; Systemic: fever, malaise, shivering/chills, fatigue, headache, sweating, myalgia, arthralgia, respiratory symptoms and diarrhoea.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes